CLINICAL TRIAL: NCT01771432
Title: Antibiotic Treatment Versus no Therapy in Kidney Transplant Recipients With Asymptomatic Bacteriuria. A Prospective Randomized Study.
Brief Title: Antibiotic Treatment Versus no Therapy in Kidney Transplant Recipients With Asymptomatic Bacteriuria
Acronym: BAC01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Núria Sabé Fernàndez (Other)
Responsible Party: Sponsor-Investigator, Núria Sabé Fernàndez, Infectious Diseases Phisycian, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FIS11-1540
Record Dates: First submitted 2012-12-21; First posted 2013-01-18 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Asymptomatic Bacteriuria; Pyelonephritis
MeSH Terms: conditions — Pyelonephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antibiotic treatment (Active Comparator): Kidney transplant recipients with asymptomatic bacteriuria will be treated with antibiotics.
  Interventions: Drug: Antibiotic treatment
- No treatment (Other): Kidney transplant recipients with asymptomatic bacteriuria will be followed without antibiotic therapy
  Interventions: Other: No treatment

INTERVENTIONS:
Drug: Antibiotic treatment — Kidney transplant recipients with asymptomatic bacteriuria will be treated with antibiotics
  Arms: Antibiotic treatment
Other: No treatment — Kidney transplant recipients with asymptomatic bacteriuria will be followed without antibiotic therapy
  Arms: No treatment

SUMMARY:
Objective: To determine whether antibiotic treatment of asymptomatic bacteriuria in kidney transplant recipients could be useful to prevent pyelonephritis in these patients.

DETAILED DESCRIPTION:
Design: Randomized prospective study. Setting: University Hospital with an active kidney transplantation program. Patients: Adult kidney transplant recipients. Interventions: Kidney transplant recipients with asymptomatic bacteriuria will be randomly assigned to be treated with antibiotics or to be followed without antibiotic therapy.

Measurements: Urine cultures will be collected weekly during the first month after transplantation, every 2 weeks until three months after transplantation, every month until 6 months after transplantation and every 3 months until 12 months after transplantation. Urine culture will be as well collected if urinary symptoms appeared.

Primary end points: To determine in both groups: the incidence of pyelonephritis.

Secondary end points: To determine outcomes in both groups (renal function, hospitalization, rejection, graft loss, opportunistic infections and mortality) and infection by multiresistant microorganisms.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive a transplant allograft during study period

Exclusion Criteria:

* No acceptation of study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
To determine the incidence of pyelonephritis in both groups | First year after kidney transplantation

SECONDARY OUTCOMES:
Renal function | First year after kydney transplantation
Need for hospitalization | First year after kydney transplantation
Incidence of graft loss | First year after kidney transplantation
Mortality | First year after kidney transplantation

OTHER OUTCOMES:
Infection by multiresistant microorganisms | First year after kydney transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Núria Sabé Fernàndez, Principal Investigator — Hospital Universitari de Bellvitge
Locations (2):
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona